CLINICAL TRIAL: NCT03462953
Title: Localization of Indicators for Epithelial Mesenchymal Transformation in Gingiva From Chronic Periodontitis Patients as Compared to Healthy Individuals (Case Control Study)
Brief Title: Identification of EMT Indicators in Healthy and Periodontally Diseased Gingival Samples
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karim wasfi wadiea, Instructor at oral biology department at Mti university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CEBC-CU-2018-02-28
Record Dates: First submitted 2018-03-04; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- individuals with healthy gingiva (Placebo Comparator): Gingival tissue samples will be harvested during the premolar extraction (Orthodontic ttt) or third molar extraction for the healthy controls.
  Interventions: Procedure: Gingival tissue samples will be harvested
- periodontally diseased individuals (Placebo Comparator): Gingival tissue samples will be harvested during periodontal surgery and extraction of the periodontally hopeless tooth for the periodontitis patients.
  Interventions: Procedure: Gingival tissue samples will be harvested

INTERVENTIONS:
Procedure: Gingival tissue samples will be harvested — Gingival tissue samples will be harvested during the premolar extraction (Orthodontic ttt) or third molar extraction for the healthy controls and during periodontal surgery or extraction of hopeless teeth with periodontal disease ..
  The dissected gingival samples will be washed in saline solution and fixed in 4% buffered formalin for 48 hours, dehydrated in ascending grades of ethyl alcohol, cleared in xylene and embedded in paraffin and will be subjected to the following:.
  1. Sections of 4-5 µm in thickness will be obtained, deparaffinized, rehydrated and subjected to histological staining and histomorphometric analysis.
  2. Real time- PCR for TGF-B1 ,Vimenten , E-Cadherin .

SUMMARY:
The current study focuses on the localization and quantitative assessment of growth factors and cytokines related to the EMT process found in the human gingival tissue samples taken from periodontally diseased individuals compared to other samples taken from healthy individuals. Through this investigation the correlation between the severity of the disease and the amount of these factors will be studied aiming to alleviation of the high prevalence of periodontal diseases among the Egyptian population.

DETAILED DESCRIPTION:
In a case control human study The existence and the amount of the indicators and cytokines for EMT in the gingival tissue samples taken from the periodontitis patients will be investigated and compared to those in healthy individuals using histopathology and real time PCR to reveal the role of these factors in periodontal disease incidence in humans.

Total of 36 participants will be recruited in this study The participants will be divided according to their periodontal status into four groups (healthy, mild, moderate and severe periodontitis) 9 patients in each group.

The periodontal screening of patients will be done using mouth mirror and graduated Williams's periodontal probe for the following:

* Gingival status will be assessed by using gingival index
* Periodontal pocket depth.
* Clinical attachment loss.
* Radiographic examination using panoramic technique. Screening criteria for chronic periodontitis was the presence of at least 5 sites with 4 mm horizontal alveolar bone loss on radiographs.

Gingival tissue samples will be harvested during periodontal surgery and extraction of the periodontally hopeless tooth for the periodontitis patients and during the premolar extraction (Orthodontic ttt) or third molar extraction for the healthy controls.

The dissected gingival samples will be washed in saline solution and fixed in 4% buffered formalin for 48 hours, dehydrated in ascending grades of ethyl alcohol, cleared in xylene and embedded in paraffin and will be subjected to the following:.

1. Sections of 4-5 µm in thickness will be obtained, deparaffinized, rehydrated and subjected to histological staining and histomorphometric analysis.
2. Real time- PCR for TGF-B1 ,Vimenten , E-Cadherin .

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for healthy group:

  * Absence of any clinical sign of gingival inflammation
  * Probing depth ≤3 mm
  * No clinical attachment loss.

Inclusion criteria for periodontitis group:

* Generalized presence of clinical signs of gingival inflammation
* Generalized probing depth ≥4 mm
* Generalized clinical attachment loss of ≥2 mm.

Exclusion Criteria:

* • Patients with any systemic disease,

  * Smokers
  * Pregnant or lactating women,
  * Cervical/proximal/subgingival caries or restorations,
  * Periodontal or antimicrobial therapy within 3 months before sampling.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-04-15 (Estimated); Primary Completion 2018-08-15 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
Localization of EMT indicators TGF- β1, Vimenten, E-Cadherin | one year
  using real time PCR the EMT indicators will be identified and quantified in all the gingival samples taken from patients of both arms of the study